CLINICAL TRIAL: NCT03731000
Title: Study of PHIL® Embolic System in the Treatment of Intracranial Dural Arteriovenous Fistulas in the Pediatric Population
Brief Title: PHIL® Embolic System Pediatric IDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alejandro Berenstein (Other)
Responsible Party: Sponsor-Investigator, Alejandro Berenstein, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 18-1298
Record Dates: First submitted 2018-08-29; First posted 2018-11-05 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2024-11

CONDITIONS: Arterio-venous Fistula; Intracranial Arteriovenous Malformations
Keywords: Pediatric
MeSH Terms: conditions — Arteriovenous Fistula; Intracranial Arteriovenous Malformations

STUDY DESIGN:
Intervention Model Description: Single Group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- PHIL® device (Experimental): Using device
  Interventions: Device: PHIL® device

INTERVENTIONS:
Device: PHIL® device — Using PHIL® device for treatment of intracranial dural arteriovenous fistulas

SUMMARY:
The purpose of this study is to collect information about how the PHIL® Embolic System works in the treatment of intracranial dural arteriovenous fistulas. Data collected in this study will be used to evaluate the safety and probable benefits in treating DAVFs.

The PHIL® Embolic System is a Humanitarian Use Device (HUD). The U.S. Food and Drug Administration (FDA) approved the use of the PHIL Embolic System as a HUD in June 2016.

DETAILED DESCRIPTION:
Study design:The study is a prospective, single-center, single-arm, clinical study evaluating outcomes in pediatric subjects with intracranial dural arteriovenous fistulas treated with PHIL® device.

Study purpose: To evaluate the safety and probable benefit of MicroVention, Inc. PHIL® Liquid Embolic material in the treatment of intracranial dural arteriovenous fistulas, alone or as an adjunctive treatment for dAVFs.

ELIGIBILITY:
Inclusion Criteria:

* Subject is <22 years of age
* Subject and legally authorized representative are willing and capable of complying with all study protocol requirements, including specified follow-up period.
* Subject's legally authorized representative(s) must sign and date an IRB approved written informed consent prior to initiation of any study procedure
* Subject has an intracranial dAVF that is deemed appropriate for embolization with PHIL without significantly increased risk to collateral or adjacent territories, OR subject has been previously treated with other embolic materials for dAVF.

Exclusion Criteria:

* Subject presents with an intracranial mass or is currently undergoing radiation therapy for carcinoma or sarcoma of the head or neck region
* Subject has known allergies to DMSO (dimethyl sulfoxide), iodine or heparin.
* Subject with a history of life threatening allergy to contrast media (unless treatment for allergy is tolerated).
* Female subject is currently pregnant.
* Subject has an acute or chronic life-threatening illness other than the neurological disease to be treated in this study including but not limited to any malignancy or debilitating autoimmune disease
* Subject has existing severe or advanced comorbid conditions which significantly increase general anesthesia and/ or surgical risk
* Evidence of active infection at the time of treatment.
* Subject has a history of bleeding diathesis or coagulopathy, international normalized ratio (INR) greater than 1.5, or will refuse blood transfusions.
* Subject weighs ≤ 2.5kg Angiographic
* Subject has severe calcification or vascular tortuosity that may preclude the safe introduction of the sheath, guiding catheter, or access to the lesion with the microcatheter.
* Contra-indication to DSA, CT scan or MRI/ MRA
* History of intracranial vasospasm not responsive to medical therapy
* Extra-cranial stenosis or parent vessel stenosis > 50% proximal to the target lesion to be treated.
* Subject has a propensity to contrast induced renal injury or a potential to nephrogenic systemic fibrosis

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-04-16 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with neurological death or major ipsilateral stroke | 12 months
  The proportion of subjects with neurological death or major ipsilateral stroke (defined as a major stroke within the vascular distribution of the vessel targeted for treatment) within 12 months following completion of treatment, reported as one composite data variable
Proportion of participants with angiographic occlusion | up to 12 months
  Proportion of subjects with Angiographic occlusion of the pre-specified target vessel intended for treatment at procedure following completion of treatment

SECONDARY OUTCOMES:
Incidence of angiographic cure | up to 12 months
  Angiographic cure of the target dAVF, defined as complete obliteration of dAVF flow following final treatment.
Incidence of new-onset permanent morbidity | up to 12 months
  New-onset permanent morbidity up to 12 month follow-up
Incidence of new-onset Intracranial hemorrhage (ICH) | up to 12 months
  New-onset Intracranial hemorrhage (ICH) up to 12 month follow0up
Number of significant technical events | up to 12 months
  Clinically significant technical events during the PHIL embolization procedure(s) including but not limited to reflux of embolic material, migration of the embolic material, catheter entrapment or damage, and vessel dissection.
Incidence of device-related adverse events at procedure | Day 1 during procedure
  Incidence of device-related adverse events at procedure at Day 1
Incidence of device-related adverse events at 30 days | at 30 days
  Incidence of device-related adverse events at 30 days.
Incidence of device-related mortality | at 30 days
  Device-related mortality at 30 days
Incidence of procedure related adverse events | up to 12 months
  Procedure related adverse events including complications of arterial puncture, contrast-induced nephropathy, renal and anesthesia-related complications.
Incidence of cranial neuropathy | up to 12 months
  Incidence of cranial neuropathy up to 12 months follow-up
Pediatric NIH Stroke Scale (PedNIHSS) | at 12 months
  PedNIHSS - 11 item instrument measuring levels of impairment on a scale of 0-42 with higher score demonstrating higher levels of impairment
The Pediatric Stroke Outcome Measure (PSOM) | at 12 months
  PSOM - measures stroke outcomes across 115 test items. On completion of the PSOM examination, the neurologist scores a Summary of Impressions containing 5 subscales: right sensorimotor, left sensorimotor (each with subcategories), language production, language comprehension, and cognitive/behavioral. Subscale scoring is 0 (no deficit), 0.5 (mild deficit, normal function), 1 (moderate deficit, decreased function), or 2 (severe deficit, missing function). The PSOM total score is the sum of the 5 subscale scores and ranges from 0 (no deficit) to 10 (maximum deficit).
Number of procedures | up to 6 months
  Number of procedures required to treat the fistula at 3-6 month follow-up
Procedure time | average of 3-4 hours
  Procedure time (defined as first to last fluoroscopic or digital subtraction angiographic acquisitions)
Dosage of Radiation exposure | average of 60 minutes
Radiation exposure time | average of 60 minutes
Injected volume of PHIL | at time of procedure, average of 3-4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Berenstein, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Tomoyoshi Shigematsu, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No